CLINICAL TRIAL: NCT02726178
Title: Cardio-respiratory Events and Inflammatory Response After Primary Immunization in Preterm Infants < 32 Weeks Gestational Age: A Randomized Controlled Study
Brief Title: Cardio-respiratory Events and Inflammatory Response After Primary Immunization in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Principal Investigator, Anne-Monique NUYT, Neonatalogist, MD, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2917
Record Dates: First submitted 2015-10-20; First posted 2016-04-01 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Complication Due to Immunization
Keywords: Apnea; bradycardia; immunization; inflammation; preterms
MeSH Terms: conditions — Apnea; Bradycardia; Inflammation | interventions — Ibuprofen; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advil® Pediatric drops for infants (Experimental): Oral ibuprofen (Advil® Pediatric drops for infants less than 3 months of age; Wyeth-Ayerst 40 mg/ml, DIN 2242522), at a dosage of 5 mg/kg/dose.
  The drug was administered 30 minutes prior to immunization, and then at 8 and 16 hours following the immunization for a total of 3 doses.
  Interventions: Drug: Advil® Pediatric drops for infants
- Control (Placebo Comparator): Oral placebo: composed of sodium stearate 0.25g + lactose 0.5g + 15 ml of simple syrup, with a measured osmolarity of about 750 mosml/kg.
  The drug (or placebo) was administered 30 minutes prior to immunization, and then at 8 and 16 hours following the immunization for a total of 3 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Advil® Pediatric drops for infants — Study the effect of inhibition of prostaglandins with ibuprofen vs placebo administration on cardio respiratory events in preterms infants
  Other Names: Oral Ibuprofen
  Arms: Advil® Pediatric drops for infants
Drug: Placebo — Study the effect of inhibition of prostaglandins with ibuprofen vs placebo administration on cardio respiratory events in preterms infants
  Other Names: Oral placebo:sodium stearate 0.25g+lactose 0.5g+15 ml syrup
  Arms: Control

SUMMARY:
Background: Inflammation may depress respiration in neonates. The aim of this study was to establish a link between post-immunization inflammation and cardio-respiratory events (CRE).

Methods: Randomized double-blind controlled study of infants born <32 weeks gestation receiving the 2 months vaccine. Infants were randomized into an ibuprofen treatment group and a placebo control group. C-reactive protein (CRP) and prostaglandins E2 (PgE2) levels were assessed before and after immunization. CRE were recorded for 72 hours. Heart rate variability (HRV) was assessed by polysomnography.

DETAILED DESCRIPTION:
Background: Immunization with the pentavalent vaccine Diphtheria-Tetanus-Acellular pertussis-Inactivated poliomyelitis-Haemophilus influenzae type b (DTPa-IPV-Hib) at two months of age is known to be associated with cardio-respiratory events (CRE), such as apnea and bradycardia, in 11 to 47% of preterm infants [1,2]

Methods: This randomized, double blinded, placebo-controlled study was conducted in the neonatal intensive care unit of Sainte-Justine University Hospital (Montreal, QC, Canada) over a period of fourteen months (February 2010 - March 2011). Study was approved by CHU Sainte-Justine institutional Ethics Committee for Clinical Studies. Written informed parental consent was obtained for all infants.

The vaccines administered were: Diphtheria-Tetanus-Acellular pertussis-Inactivated polio-Haemophilus influenzae type B (DTaP-IPV-HIB: Pediacel® 0.5ml) and the pneumococcal conjugate 10-valent vaccine (Synflorix® 0.5ml). The two vaccines were administered by nurses intramuscularly in the anterolateral region of each thigh.

On enrollment, patients were randomized by the pharmacy (investigator blinded) into two groups: the study group received oral ibuprofen (Advil® Pediatric drops for infants < 3 months of age; Wyeth-Ayerst 40 mg/ml, DIN 2242522) 5 mg/kg/dose as recommended by the manufacturer (Ibuprofen; n=28):http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails.

The control group received an oral placebo (Placebo; n=28). The placebo was prepared by the CHU Sainte-Justine pharmacy and was composed of sodium stearate 0.25g + lactose 0.5g + 15 ml of simple syrup, with a measured osmolarity of about 750 mosml/kg. The drugs were administered by nurses in an opaque syringe 30 minutes prior to immunization, and then at 8 and 16 hours following the immunization for a total of 3 doses.

Cardio-respiratory monitoring and recordings were performed in all patients continuously for 72 hours, beginning 24 hours before and continuing until 48 hours after immunization (Figure 1). Monitoring tracings were printed and CRE were extracted and compared to nurses' surveillance noted in a separate sheet. These analyses were performed by two different operators: a medical fellow (WBJ) and a research nurse. The results were discussed and an agreement reached between operators in any instances of discordance. The recorded CRE included: bradycardia (a 33% decrease in baseline heart rate for at least 4 seconds or a heart rate ≤ 80 bpm), desaturations (10% decrease in baseline saturation), and apnea (respiratory pause of at least 20 seconds, or a respiratory pause of 15 seconds associated with a bradycardia).

Total CRE was expressed as the average number of events (desaturation + apneas + bradycardia) / 24 hours. Δ Total CRE / patient / 24 hours was defined as the difference between the average number of events / 24 hours observed before vs. after immunization for each patient. Biographical data, maternal and pregnancy data, and infant medical data (base line heart rate, temperature and ventilation duration) were also collected for each patient.

Two annotated polysomnographies were performed for all patients with an AURA PSG GRASS ambulatory and wireless system. Each polysomnography had a duration of 2.5 hours: the first was conducted on enrolment (the day before immunization), and the second was conducted 18 to 24 hours after immunization. The patients were settled comfortably in an environment with reduced tactile, auditory and luminous stimulation, and the cardiac electrodes, oximeter and abdominal respiration detector were placed. The polysomnographies were annotated by the research nurse or medical fellow (WBJ) for the total duration of the recordings, and analysis was performed by the team of Pr Pladys (Rennes, France).

CRP and prostaglandin E2 were measured as systemic markers of inflammation. Blood samples for CRP levels were taken at the same time (0.5ml/sample in microtube with lithium heparin and gel barrier), and analyzed by immunoturbidimetric dosage (Sainte-Justine University Hospital Biochemistry laboratory). Capillary blood samples (0.5ml/sample) were collected in an EDTA-coated tube 30-60 min prior to the immunization, and 18h after. 10µM indomethacin was added to each tube within 30 min of sampling in order to inhibit ongoing PG synthesis by platelets. After centrifugation, plasma was frozen (-80ºC) until analysis. Plasma PGE2 concentration was determined by ELISA (PGE2 Parameter Assay kit; R and D systems, #KGE004B; intra- and inter-assay variability of 6.7% and 10.6% respectively).

All blood samples were taken following sucrose administration as per routine practice in the NICU. They also were taken at the same time of a routine blood test already planned for the patients. Δ CRP and Δ PGE2 were defined, respectively, as the difference between CRP and PGE2 levels before and after immunization.

Statistical analysis was performed using SPSS (v20.0 for Windows). All variables were tested for normal distribution using the Shapiro-Wilk normality test. When normally distributed (parametric), data were presented as mean ± standard deviation, applying one-way analysis of variance (ANOVA) and Bonferroni post hoc test. Nonparametric data were analyzed using the Kruskall-Wallis with Dunn post-test. HRV parameters were analyzed by paired or unpaired Student's t-test, or Wilcoxon w-test and Mann-Whitney u-test as appropriate. Correlations between non parametric data were analyzed using Spearmen test. The two-sided significance level was set at 0.05.

The sample size calculation (26 patients required in each group) was based on a 40% incidence of CRE post vaccination [1,2] and with the hypothesis that the ibuprofen will decrease this incidence from 40% to 15% (α of 0.05 and a power of 80%).

A post-hoc analysis was performed to identify the pre-immunization characteristics of the preterm infants who increased their CRE of more than 1 SD.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants less than 32 weeks of gestational age
* Postnatal age more than 7 weeks
* Informed parental consent

Exclusion Criteria:

* anomalies in cardiac conduction
* congenital malformations
* severe intraventricular haemorrhage (grade 3 or 4) or with periventricular leukomalacia

Min Age: 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Monique Nuyt, MD, Principal Investigator — Ste-Justine's hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoch B, Bernhard M. Central apnoea and endogenous prostaglandins in neonates. Acta Paediatr. 2000 Nov;89(11):1364-8. doi: 10.1080/080352500300002589. PMID 11106051
- [Background] Schulzke S, Heininger U, Lucking-Famira M, Fahnenstich H. Apnoea and bradycardia in preterm infants following immunisation with pentavalent or hexavalent vaccines. Eur J Pediatr. 2005 Jul;164(7):432-5. doi: 10.1007/s00431-005-1674-3. Epub 2005 Apr 21. PMID 15843978
- See also: the full bibliographic citation of the article on Pubmed — https://www.ncbi.nlm.nih.gov/pubmed/?term=Cardio-respiratory+Events+and+Inflammatory+Response+After+Primary+Immunization+in+Preterm+Infants+%3C+32+Weeks+Gestational+Age%3A+A+Randomized+Controlled+Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process was conducted in the neonatal intensive care unit of Sainte-Justine University Hospital (CHU Sainte-Justine, Montreal, QC, Canada) over a period of fourteen months (February 2010 - March 2011).
Pre-assignment Details: A total of 362 preterm infants were screened, 56 completed the study. Of the infants who did not participate in the study, 212 were discharged before the first immunization (92 to home and 120 to level II nurseries), 37 died, 28 were still intubated at the time of enrolment, 14 did not meet the inclusion criteria, and parents refused for 15.
Groups:
- Advil® Pediatric Drops for Infants: Oral ibuprofen (Advil® Pediatric drops for infants less than 3 months of age; Wyeth-Ayerst 40 mg/ml, DIN 2242522), at a dosage of 5 mg/kg/dose.
  The drug was administered 30 minutes prior to immunization, and then at 8 and 16 hours following the immunization for a total of 3 doses.
  Advil® Pediatric drops for infants: Study the effect of inhibition of prostaglandins with ibuprofen vs placebo administration on cardio respiratory events in preterms infants
- Control: Oral placebo: composed of sodium stearate 0.25g + lactose 0.5g + 15 ml of simple syrup, with a measured osmolarity of about 750 mosml/kg.
  The drug (or placebo) was administered 30 minutes prior to immunization, and then at 8 and 16 hours following the immunization for a total of 3 doses.
  Placebo: Study the effect of inhibition of prostaglandins with ibuprofen vs placebo administration on cardio respiratory events in preterms infants
Period: Overall Study
Arm/Group | Advil® Pediatric Drops for Infants | Control
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advil® Pediatric Drops for Infants | Control | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 27.8 (1.8) | 27.2 (2) | 27.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Number of CRE (Extracted From Printed Monitoring Tracings Compared to Noted Nurses' Surveillance) Following the First Dose of Pentavalent Vaccine in Preterm Infants Born < 32 Weeks Gestation After Administration of Ibuprofen.
Description: Immunization with the pentavalent vaccine Diphtheria-Tetanus-Acellular pertussis-Inactivated poliomyelitis-Haemophilus influenzae type b (DTPa-IPV-Hib) at two months of age is known to be associated with cardio-respiratory events (CRE), in 11 to 47% of preterm infants.It is considered that the immature brainstem respiratory control of preterms make them more vulnerable to the inflammatory reaction caused by immunization. We hypothesized that post-immunization CRE are correlated with inflammatory reaction. The primary objective was to examine the impact of endogenous PG inhibition on the occurrence of CRE following the first dose of pentavalent vaccine in preterm infants born < 32 weeks gestation. Total CRE was expressed as the average number of events (desaturation + apneas + bradycardia) / 24 hours. Δ Total CRE / patient / 24 hours was defined as the difference between the average number of events / 24 hours observed before vs. after immunization for each patient.
Time Frame: the mean of CRE occured in the 48h after immunization minus the base line CRE : mesured 24h before immunization
Measure: Mean (Standard Deviation); unit: events/patient/24hours
Arm/Group | Advil® Pediatric Drops for Infants | Control
Number analyzed (Participants) | 28 | 28
events/patient/24hours | 0.1 (8) | 5.4 (10)

2. Secondary Outcome: The Modifications in HRV That Can Predict the Occurrence of CRE in Preterm Infants After Immunization.
Description: The secondary objective was to identify predictive factors of occurrence of CRE in preterm infants after immunization through the analysis of their HRV. Two annotated polysomnographies were performed for all patients with an AURA PSG GRASS ambulatory and wireless system. Each polysomnography had a duration of 2.5 hours: the first was conducted on enrolment (the day before immunization), and the second was conducted 18 to 24 hours after immunization : we compared the mean of the datas of polysomnographies after to those before immunization.
Time Frame: 72 h
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Advil® Pediatric Drops for Infants; Control: Two annotated polysomnographies were performed for all patients:
  The first annotated polysomnography was conducted the day before immunization and had a duration of 2.5 hours.
  The second was conducted 18 to 24 hours after immunization.
  We compared the data of polysomnographies after to those before immunization.
  Polysomnography : an AURA PSG GRASS ambulatory and wireless system.
Arm/Group | Advil® Pediatric Drops for Infants | Control
Number analyzed (Participants) | 28 | 28
msec | -10 (36) | -8 (28)

ADVERSE EVENTS:
Time Frame: 2 days after the first immunization
Arm/Group | Advil® Pediatric Drops for Infants | Control
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

LIMITATIONS AND CAVEATS:
1-the small number of patient recruted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes